CLINICAL TRIAL: NCT05470244
Title: Effects of Transcutaneous Electrical Nerve Stimulation in Post-operative Total Knee Arthroplasty Recovery and Intra-venous Analgesics Requirement
Brief Title: TENS in Post-operative Total Knee Arthroplasty Recovery and Intra-venous Analgesics Requirement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Ayesha Jamil, Assistant Professor, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TKR
Record Dates: First submitted 2022-07-12; First posted 2022-07-22 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Total Knee Arthoplasty; Knee Pain
Keywords: Total Knee Arthoplasty; Knee Pain; Post-operative; Transcutaneous electrical nerve stimulation; Intra-venous; Analgesics requirement; Recovery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be unaware of the treatment group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Exercise Group (Active Comparator): This group will receive Routine Physical therapy protocol along with prescribed intra-venous regimen.
  Interventions: Other: Routine Physical Therapy and Intra-venous analgesic regimen
- TENS Plus Therapeutic Exercise Group (Experimental): This group will receive high frequency Transcutaneous Electrical Nerve Stimulation with routine physical therapy and prescribed intra-venous regimen.
  Interventions: Other: Transcutaneous Electrical Nerve Stimulation along with Routine Physical Therapy and Intra-venous analgesic regimen

INTERVENTIONS:
Other: Routine Physical Therapy and Intra-venous analgesic regimen — ROM Exercises will be performed and analgesics including the NSAIDs and narcotics as per prescription of surgeon/physician will be given to all subjects
  Arms: Therapeutic Exercise Group
Other: Transcutaneous Electrical Nerve Stimulation along with Routine Physical Therapy and Intra-venous analgesic regimen — High frequency stimulations via Transcutaneous Electrical Nerve Simulator will be applied. ROM Exercises will be performed and analgesics including the NSAIDs and narcotics as per prescription of surgeon/physician will be given to all subjects
  Arms: TENS Plus Therapeutic Exercise Group

SUMMARY:
Total knee arthroplasty (TKA) is among the major advancements for the treatment of knee pain and improvement of physical function when conservative management fails to comply with. The success of this arthoplasty results in more functional mobility and better quality of life. However, management of pain after TKA in post-operative period is a big challenge to deal.

DETAILED DESCRIPTION:
Transcutaneous electrical nerve stimulation is a cost effective, non-invasive electrotherapeutic modality used in alleviating pain in both acute and chronic conditions affecting neuromusculoskeletal system of the body.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female
2. Aged between 31-70 years
3. Total Knee Arthoplasty, who had been diagnosed with knee osteoarthritis, inflammatory arthritis, trauma, fracture result in total knee arthoplasty.

Exclusion Criteria:

1. Any allergic condition of skin
2. Chronic consumption of opioids
3. History of dysplasia or malignancy to knee joint
4. Any major bone operation of lower limb
5. BMI higher than 35 kg m-2
6. History of mental disorder
7. Neurological illness e.g. Alzheimer which might interfere with assessment process.

Ages: 31 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | Pain intensity will be measured at baseline,and change in pain intensity will be measured from baseline to 24 hour, 48 hour and 72 hours.
  Pain intensity will be measured using Visual Analogue Scale
Rang of Motion | Knee Range of Motion will be measured at baseline, and Change in Knee Range of Motion will be measured from baseline to 24 hour, 48 hour and 72 hours
  Knee Rang of Motion will be measured using Universal Goniometer
Intra-venous analgesic requirement | Analgesics requirement will be observed at first post-operative day, at second post-operative day, at third post-operative day
  Dose and frequency of intravenous analgesic requirement will be observed through Patient's file

SECONDARY OUTCOMES:
Length of Hospital Stay | It will be measured from the time of randomization till the time of discharge from hospital upto ten days
  Length of Hospital Stay of patient

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Ashfaq Ahmed, PhD, Study Director — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
it will be shared immediately after publication
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending on 36th month